CLINICAL TRIAL: NCT06713655
Title: Multicenter Study on PAX1 Methylation for Predicting Lesion Persistence/Recurrence in HSIL Patients with Positive Margins After Cervical Conization
Brief Title: Predicting Treatment Failure in HSIL Patients with Positive Margins After Conization Via Detection of PAX1 Methylation
Status: Not yet recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Huzhou Maternity and Child Care Hospital (Unknown); Jiaxing Maternity and Child Health Care Hospital (Other); Shaoxing Maternity and Child Health Care Hospital (Other); Ningbo No. 1 Hospital (Other); Jinhua Central Hospital (Other); Taizhou Hospital Zhejiang Province (Unknown)
Responsible Party: Principal Investigator, Weiguo Lv, Professor, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: IRB-20240248-R
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: High-grade Squamous Intraepithelial Lesions (HSIL); Cervical Conization
Keywords: cervical intraepithelial neoplasia; conization; positive margins; cervical cancer; treatment failure; residual/recurrent disease
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Uterine Cervical Dysplasia; Margins of Excision; Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this multicenter, observational study is to evaluate whether methylation testing of paired box gene 1 (PAX1) can better predict and diagnose recurrence or persistent disease in patients with positive margins after cervical conization for high-grade squamous intraepithelial lesion (HSIL). The main question it aims to answer is:

Can PAX1 gene methylation testing provide a more accurate and effective prediction and diagnosis of cervical disease recurrence/persistence in addition to existing methods? Participants will be managed according to the latest clinical guidelines, and during follow-up, a non-invasive test, PAX1 gene methylation testing, will be added.

DETAILED DESCRIPTION:
This study is a multicenter, prospective observational study that qualitatively assesses the methylation status of the PAX1 gene in cervical exfoliated cells from patients with HSIL and positive margins after conization. The aim is to evaluate the ability of PAX1 gene methylation testing to predict treatment failure (lesion recurrence or persistence). The first follow-up occurs 6 months post-surgery, including high-risk human papillomavirus (hrHPV) testing and cytology, with referral for colposcopy, including biopsy and/or endocervical curettage (ECC), if necessary. Subsequent management and follow-up are based on examination results, following clinical guidelines, and arranged at intervals of 6-12 months depending on the findings. The follow-up includes routine clinical examinations widely applied in practice, and PAX1 testing will be completed at each follow-up visit. PAX1 testing, like hrHPV testing and cytology, will be performed using cervical exfoliated cells.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 25 years and less than 55 years;
* First-time cervical conization (cold knife conization or loop electrosurgical excision procedure);
* Postoperative pathology showing HSIL (CIN2 or CIN3);
* Positive margins for HSIL (CIN2 or CIN3) in conization specimen.

Exclusion Criteria:

* The presence of other malignant tumors or precancerous lesions;
* Lack of willingness for follow-up;
* Pregnant or breastfeeding women;
* Unable or unwilling to complete follow-up examinations;
* History of prior cervical disease treatment (surgical or physical therapy);
* Presence of immune system disorders.

Ages: 26 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing their first cervical conization surgery for treatment or diagnosis at seven hospitals mentioned above in Zhejiang Province.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate within 24 months after surgery (cervical intraepithelial neoplasia grade 2+ (CIN2+) recurrence/residual rates) | 2 years post-surgery
  the percentage of HSIL treatment failure (CIN2+ recurrence and residual) within 24 months after surgery
Sensitivity of the PAX1 methylation to detect treatment failure | 2 years post-surgery
specificity of the PAX1 methylation to detect treatment failure | 2 years post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No